CLINICAL TRIAL: NCT04207918
Title: A Phase II Study of Chemoradiotherapy With Nimotuzumab in Unresectable Esophageal Squamous Cell Carcinoma Based on Nutritional Risk Screening Score (NRS2002)
Brief Title: A Phase II Study of Chemoradiotherapy With Nimotuzumab in Unresectable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/291-2075
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer; Chemoradiotherapy; Nimotuzumab; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; nimotuzumab; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemoradiotherapy（NCRT） (Experimental): NCRT arm receives intensity-modulated radiotherapy concurrently with S-1（40-60/m2/d，orally twice a day） and nimotuzumab（400mg/d，by intravenous infusion once a week）.
  Interventions: Radiation: Radiotherapy; Drug: Nimotuzumab; Drug: S-1

INTERVENTIONS:
Radiation: Radiotherapy — 44.94Gy and 37.8Gy in 21 fractions to PGTV and PTV for neoadjuvant treatment. 59.92Gy and 50.4Gy in 28 fractions to PGTV and PTV for definitive treatment.
Drug: Nimotuzumab — 400mg, by intravenous infusion once a week in 4-6 weeks.
Drug: S-1 — 40-60mg/m2/d，orally twice a day concurrently with radiotherapy.

SUMMARY:
This phase II clinical study is designed to evaluate the 1 year local tumor control rates after the targeted therapy of intensity-modulated radiation therapy synchronized chemotherapy with nimotuzumab combined with S-1 in local advanced esophageal squamous cell carcinomas based on Nutritional Risk Screening NRS2002.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Pathologically or cytologically proven esophageal squamous cell carcinomas in patients staged as T2-4N0-1M0-1b (AJCC 6th TNM staging, M1b limited to clavicular or celiac lymph node metastasis)
* Primary treatment accepted in Chinese Academy of Medical Sciences
* KPS ≥70
* NRS score ≥2
* Cervical or thoracic esophageal cancer histologically proved esophageal cell carcinoma
* Normal organ and marrow function as defined below:

Hemoglobin: greater than or equal to 100g/L ;Leukocytes: greater than or equal to 3,500 G/L; Neutrophil: greater than or equal to 1,500 G/L; Platelets: greater than or equal to 100,000/mm3 ; Creatinine within normal upper limits; BUN within normal upper limits; AST/ALT: less than or equal to 1.5 times the upper limit; Total bilirubin: less than or equal to 1.5 times the upper limit; Alkaline phosphatase :less than or equal to 1.5 times the upper limit

* Informed consent

Exclusion Criteria:

* Patients with other cancer history in 5 years except cervical carcinoma in situ and non-malignant melanoma skin cancer
* Any prior chemotherapy or other cancer treatment prior to this protocol
* With any distant metastasis in liver, lung, bone, CNS or peritoneal transplantation
* History of allergic reactions attributed to contrast medium, similar chemical or biologic complex
* Existing esophageal fistula, perforation and cachexia
* Existing active infection such as active tuberculosis and hepatitis
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* Participation in other clinical trials currently or within 4 weeks of selection
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Local control rate | 1 year

SECONDARY OUTCOMES:
Number of Participants with acute toxicities | 2-3 months
  Acute toxicities are evaluated by NCI-CTC version 5.0
R0 resection rate | 2-3 months
  The surgical procedure was radical esophagectomy after neoadjuvant therapy.
Pathological response rate | 2-3 months
  Pathological response were classified into five grades according to Mandard Tumor Regression Grade.
Tumor Response rate | 2-3 months
Incidence of perioperative complications | 2-3 months
  During hospital stay and within the first 30 days after completion of surgery.
Overall survival | 1 year, 2 year
Progression free survival | 1 year, 2 year
Texture analysis of CT and/or MRI simulation in predicting tumor response rate and prognosis | 1 year, 2 year
ctDNA in predicting tumor response rate and prognosis | 1 year, 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China